CLINICAL TRIAL: NCT07015112
Title: Applying a Multidisciplinary Intervention for Drug Adequacy in a Intermediate Care Hospital (AMIDA-ICH)
Brief Title: Applying a Multidisciplinary Intervention for Drug Adequacy in an Intermediate Care Hospital (AMIDA-ICH)
Acronym: AMIDA-ICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc Sanitari Pere Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMIDA-ICH
Record Dates: First submitted 2025-06-01; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Poly Pharmacy; Frail Elderly
Keywords: polypharmacy; frailty; adverse drug event; deprescribing
MeSH Terms: conditions — Frailty; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Stepped-wedge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (usual care) (No Intervention): Control arm will receive usual standard of care
- Intervention (patient-centered medication review) (Experimental): Intervention arm will receive a multidisciplinary patient-centered medication review
  Interventions: Other: Patient-centered multidisciplinary treatment review

INTERVENTIONS:
Other: Patient-centered multidisciplinary treatment review — Patient-centered multidisciplinary treatment review is defined as a medication review conducted by a multidisciplinary team (geriatrician, clinical pharmacist, nurse) according to a patient-centered methodology, based on person-centered evaluation of both personal and clinical insights, diagnostic-centered evaluation (based on current guidelines), and drug-centered evaluation (based on adequacy)
  Arms: Intervention (patient-centered medication review)

SUMMARY:
The goal of this clinical trial is to learn if a multi-professional (conducted by geriatricians, clinical pharmacists, nurses) medication revision, centered on patients' goals and characteristics, can improve treatment adequacy in older adults admitted to an intermediate care hospital.

The main question it aims to answer is: does this approach reduce the average number of medications taken per patient?

Researchers will compare this multi-professional patient-centered revision to the usual standard of care (treatment revision conducted by a clinical pharmacist) to see if the patient-centered revision works in improving treatment adequacy.

Participants admitted to an intermediate care hospital will undergo a comprehensive assessment by a geriatrician, and a medication revision (conducted by a multidisciplinary team or a clinical-pharmacist alone). They will also be asked to fulfill some questionnaires on their health status and attitudes. Any possible adverse events to the medications will be recorded at discharge. Participants will be contacted again three months after discharge to check for any readmission or death.

ELIGIBILITY:
Inclusion Criteria:

* older adults (65+ years)
* ≥ 3 or more chronic conditions requiring medical therapy
* able to speak Spanish
* capacity to provide informed consent or have a surrogate able to consent on their behalf

Exclusion Criteria:

* unable to provide informed consent
* anticipated length of hospital stay < 72h
* estimated life expectancy < 3 months
* homeless
* already enrolled in a drug trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of drugs | Baseline and after discharge, an average of 30 days
  Median number of drugs per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Parc Sanitari Pere Virgili, Barcelona, Barcelona, Spain